CLINICAL TRIAL: NCT01235702
Title: Multiple CVD Risk Reduction in Adult African-Americans: A Pilot Study
Brief Title: Metro Atlanta Heart Disease Study - II (MAHDS II)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Sharon K Davis, PhD Director- Social Epidemiology Research Center, Morehouse School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TS-0724
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2003-03

CONDITIONS: African Americans With Hypertension.
Keywords: high blood pressure, hypertension, African Americans, perceived stress
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 12-week lifestyle modification

SUMMARY:
A 12-week treatment/control trial was implemented to assess the effects of a multi component lifestyle program on improvements in body mass index, weight, perceived stress and blood pressure in African American men and women who were at increased risk for cardiovascular disease. It was hypothesized that treatment group would experience significant improvements when compared to the control group.

ELIGIBILITY:
Inclusion Criteria: African American men and women aged >21 with elevated blood pressure and excess body weight who resided in metro Atlanta, GA.

-

Exclusion Criteria: Individuals with normal blood pressure and body weight, as well as those residing outside of metro Atlanta, GA. Individuals with psychological conditions were also excluded.

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2002-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
blood pressure | 10/2002 - 11/2003
  a 12-week behavior modification program was implemented to assess the effects of nutrition counseling, stress reduction education, and directed physical activity on African Americans at increased risk for cardiovascular disease.

SECONDARY OUTCOMES:
body weight | 10/2002 - 11/2003

CONTACTS AND LOCATIONS:
Overall Officials: Sharon K Davis, PhD, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States